CLINICAL TRIAL: NCT06147414
Title: Evaluation of the Diagnostic Performance of Non-Invasive Prenatal Diagnosis for Single Gene Disorders
Brief Title: Development of Non-Invasive Prenatal Diagnosis for Single Gene Disorders
Acronym: DANNIgene
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220809; 2023-A00821-44 (Other: ID-RCB)
Record Dates: First submitted 2023-09-18; First posted 2023-11-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Invasive PreNatal Diagnosis in a Context of Family History of Single-gene Disorders, Including; Sickle Cell Disease; Cystic Fibrosis; Fragile X Syndrome; Proximal Spinal Muscular Atrophy; Myotonic Dystrophy; Muscular Dystrophy, Duchenne; Muscular Dystrophy, Becker; Neurofibromatosis-Noonan Syndrome; Huntington Disease; Hemophilia A; Hemophilia B; MODY2 Diabetes; X-Linked Hydrocephalus; Autosomal Recessive Polycystic Kidney Disease
Keywords: Gene HBB; Gene CFTR; Gene FMR1; Gene SMN1; Gene DMPK; Gene DMD; Gene NF1; Gene HTT; Gene F8; Gene F9; Gene GCK; Gene L1CAM; Gene PKHD1
MeSH Terms: conditions — Anemia, Sickle Cell; Cystic Fibrosis; Fragile X Syndrome; Myotonic Dystrophy; Muscular Dystrophy, Duchenne; Neurofibromatosis-Noonan syndrome; Huntington Disease; Hemophilia A; Hemophilia B; Hydrocephalus, X-linked; Polycystic Kidney, Autosomal Recessive; Neurofibromatoses | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant women undergoing invasive PND in a context of family history of SGD: SGD-NIPD will be proposed by CPDPN recruitment centres to pregnant women undergoing invasive PND in a context of family history of SGD because of parental pathogenic mutation.s in one of the following gene: HBB, CFTR, FMR1, SMN1, DMPK, DMD, NF1, HTT, F8, F9, GCK, L1CAM, PKHD1 or ATP7A
  Interventions: Biological: Blood sample
- pregnant women undergoing prenatal counselling in a context of maternal history of diabetes MODY-GCK
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — A blood sample (50 ml) will be taken in care of prenatal diagnosis and 40 ml will be used for study.
  The 40 mL of blood needed for the research will be collected on BCT tubes (4 tubes).
  During the study, in centers, the plasma samples will be stored at room temperature and will be sent to the laboratory within 24 hours (no centrifugation in centers).
  The plasma samples will be then temporarily stored at -80°C in each co-investigating laboratory under the supervision of lab supervisor until the analysis. cfDNA will be extracted from the whole plasma sample before each sequencing run and stored à +4°C until the cfDNA sequencing.

SUMMARY:
Cell-free fetal DNA (cffDNA) is present in the maternal blood from the early first trimester of gestation and makes up 5%-20% of the total circulating cell-free DNA (cfDNA) in maternal plasma. Its presence in maternal plasma has allowed development of noninvasive prenatal diagnosis for single-gene disorders (SGD-NIPD). This can be performed from 9 weeks of amenorrhea and offers an early, safe and accurate definitive diagnosis without the miscarriage risk associated with invasive procedures. One of the major difficulties is distinguishing fetal genotype in the high background of maternal cfDNA, which leads to several technical and analytical challenges. Besides, unlike noninvasive prenatal testing for aneuploidy, NIPD for monogenic diseases represent a smaller market opportunity, and many cases must be provided on a bespoke, patient- or disease-specific basis. As a result, implementation of SGD-NIPD remained sparse, with most testing being delivered in a research setting.

The present project aims to take advantage of the unique French collaborative network to make SGD-NIPD possible for theoretically any monogenic disorder and any family.

DETAILED DESCRIPTION:
Since the identification of cffDNA in maternal plasma in 1997, there have been rapid developments in exploiting its presence for prenatal diagnosis and screening. The first proof of principle studies using cfDNA from maternal plasma to detect fetal aneuploidy were published in 2008 following which there was rapid commercialization. Nowadays, non-invasive prenatal testing (NIPT) for aneuploidies is widely used across the world as a screening test for the most frequent fetal trisomies. Unlike non-invasive prenatal testing, where a positive result requires confirmation following an invasive test, non-invasive prenatal diagnosis (NIPD) offers the advantage of a definitive diagnosis without an invasive procedure - and its associated miscarriage risk - because confined placental mosaicism does not occur with NIPD for single-gene disorders (SGD).

NIPD can be offered earlier in pregnancy than invasive testing, from 7 weeks of gestation. This can reduce parental anxiety and allows more time for decision-making and planning. Indeed, there are substantial challenges to overcome for SGD-NIPD. i/ Circulating cffDNA, which is released from the placenta from about 4 weeks gestation, makes up only 5%-20% of total circulating cfDNA in maternal plasma. This percentage increases with gestation and is influenced by factors such as maternal weight, smoking, and pregnancy complications such as preeclampsia. Consequently, optimized techniques and highly sensitive detection approaches are required to detect variants in the fetal DNA. ii/ fetal fraction must be calculated to confirm that there are sufficient levels of cffDNA present and to avoid false negative results. iii/ Another issue is the short fragment length of cffDNA, which makes detection of triplet repeats and large deletions or duplications challenging.

Besides fetal sex determination and fetal Rhesus D status, principal investigator's team was the first to propose SGD-NIPD for use in clinical practice in France for autosomal disorders caused by de novo or paternally inherited mutations, for which variants in the fetal DNA can easily be distinguished in the high background of maternal cfDNA. Droplet-digital Polymerase Chain Reaction or Next-Generation Sequencing can be used to target a single mutation for this analysis.

However, this approach requires mutation-specific developments and is restricted to point mutations that are absent from maternal DNA. NIPD for X-linked disorders, as well as autosomal dominant maternally inherited or autosomal recessive disorders for which both parents are carriers of the same mutation has posed a greater challenge. A quantitative approach is needed to ascertain fetal inheritance of the maternal mutation. In autosomal dominant diseases with maternal mutation or autosomal recessive diseases, the ratio between the total copies of the mutant allele (M) and the wildtype allele (N) in the maternal plasma contributed by both the maternal and fetal cell-free DNA is expected to be balanced (M=N) if the genotype of the fetus (M/N) is identical to the mother (M/N). However, the allelic ratio will be imbalanced if the fetal genotype is different from the maternal genotype. If the fetus has inherited both parental wildtype alleles (N/N), there would be additional dosage of the wildtype allele in the maternal plasma contributed from the fetus, resulting in under-representation in the total copies of the mutant allele (M<N). Conversely, if the fetus has inherited the parental mutant alleles (M/M), there would be additional dosage of the mutant allele in the maternal plasma contributed from the fetus, resulting in over-representation in the total copies of the mutant allele (M>N). The degree of expected allelic imbalance in maternal plasma depends on the DNA fetal fraction in the maternal plasma.

A quantitative relative mutation dosage (RMD) approach has been developed to detect such mutant allelic imbalance. This approach has been applied to the non-invasive detection of recessive disorders such as beta-thalassemia and sickle cell anemia but also for X-linked disorders like hemophilia . Nevertheless, direct interrogation of the mutation appears to be difficult - even impossible - in certain genomic loci due to the presence of repetitive sequences, homologous pseudogenes, and undefined genomic rearrangement. Moreover, successful classification of allelic imbalance is statistically dependent on the available copies of mutant and wildtype alleles in the blood sample, hampered by the very low absolute concentration of cfDNA. As a result, RMD analysis is still at a proof-of-concept phase, being evaluated in a limited number of studies, with a limited number of patients, and has never been implemented in standard care diagnosis to investigator's knowledge.

These challenges have inspired an alternative solution with indirect mutational status inference by relative haplotype dosage analysis (RHDO). SGD-NIPD by indirect mutational status inference by RHDO has been shown to be successful for -thalassemia and is now in clinical practice only in the United Kingdom National Health Service for cystic fibrosis, spinal muscular atrophy and Duchenne muscular dystrophy. Although RHDO has been proven reliable, quality controls and decisional thresholds are not thoroughly addressed for clinical implementation.

Principal investigator's team got inspired from the approach developed by Dennis Lo and enriched the methodological aspect i/ by comprehensively allowing to control the statistical errors; ii/ by distinctly identifying key parameters that influence the diagnosis performance of RHDO; iii/ by pinpointing output features illustrating the overall quality of the test.

All these factors were then merged, resulting in quality scores and decision threshold definition.

A preliminary fruitful work involving more than 90 at risk families for 5 disorders was conducted by principal investigator's team.

Altogether, the workflow appears to be:

Specific: 92/92 (100%) fetal genotype correctly identified, among conclusive tests (i.e. 92 concordant + 0 discordant results) Sensitive: 92/98 (94%) conclusive tests, among all tests (i.e. 92 conclusive concordant results + 6 inconclusive concordant results) Clinically viable: turn-around-time of 5-6 working days. Universal: applicable to any mutational profile (point mutation, deletion, duplication, triplet expansion etc.).

Adaptable: can be easily modified for testing of other SGDs. The present project aims to take advantage of the unique French collaborative network to make SGD-NIPD possible for theoretically any monogenic disorder and any family. The investigators wish to build on this preliminary work to broaden the workflow to each disease of interest for a comprehensive evaluation of the diagnostic performance of SGD-NIPD. Eventually, this collaborative achievement will allow the redraw of French landscape of prenatal diagnosis.

One advantage of the approach proposed in this study is that it is targeted. The RHDO analysis and its result will be specific of DNA locus involved in the family disorder, and will not affect other regions of the genome. Consecutively, investigators will not be confronted to ethical and social issues surrounding full exome or genome sequencing in the prenatal setting, for example the counselling issues that arise through the identification of variants of uncertain significance or incidental findings.

SGD-NIPD will be proposed by Multidisciplinary Centers for Prenatal Diagnosis to pregnant women undergoing invasive prenatal diagnosis in a context of family history of single-gene disorders because of parental pathogenic mutation.s in one of the following gene: HBB, CFTR, FMR1, SMN1, DMPK, DMD, NF1, HTT, F8, F9, GCK, L1CAM, PKHD1 or ATP7A.

In the case of MODY-GCK diabetes, fetal growth is dependent on fetal genotype. Insulin treatment should be considered to reduce the risk of macrosomia only in the 50% of MODY-GCK mothers with unaffected foetus. However, invasive PND is not recommended in clinical care due to a significant benefit/risk imbalance. For these MODY-GCK cases, the result of the SGD-NIPD will be compared to the genotype result of the newborn at birth, already planned as part of routine care. The benefits of NIPD in the pregnancy management of women with pathogenic GCK variants has been demonstrated by international experts of monogenic diabetes.

If the baby inherits the maternal GCK variant - the baby would be expected to have a normal birthweight as per background population.

Treatment of maternal hyperglycemia is not recommended in those cases as the baby would not be expected to have a higher risk of being born large-for-gestational-age than the background population.

However, if the baby does not inherit the maternal GCK variant, it would have a higher risk of macrosomia / large-for-gestational-age (~800g increase in birth weight). Monitoring of fetal growth ultrasound (28,32,36 weeks), treatment for maternal hyperglycemia with insulin, and planning delivery at 37-39 weeks gestation is recommended to try to limit fetal growth.

Recruitment capacities are assessed by considering the prevalence of rare diseases and the activities of each co-investigator center as reported annually in the report of the biomedicine agency.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman with 9 weeks of amenorrhea or more
* singleton pregnancy
* undergoing invasive PND in a context of family history of SGD involving the following genes : HBB, CFTR, FMR1, SMN1, DMPK, DMD, NF1, HTT, F8, F9, GCK, L1CAM, PKHD1, ATP7A or undergoing prenatal counselling in a context of maternal history of diabetes MODY-GCK
* germinal pathogenic paternal and/or maternal mutations previously identified
* age 18 years old or over
* signing an informed consent

Exclusion Criteria:

* at risk of SGD involving a de novo pathogenic mutation in a previous child
* woman under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant woman undergoing genetic counselling in a context of family history of SGD either through prenatal diagnosis by invasive sampling or through postnatal diagnosis by sampling of the newborn (for MODY-GCK)
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
% of affected/unaffected fetuses that were correctly classified as affected/unaffected | 1 day
  respectively among conclusive results
% of inconclusive results | 1 day

SECONDARY OUTCOMES:
cffDNA concentration in maternal plasma | 1 day
  relative concentration in % of total cell-free DNA
sequencing coverage | 1 day
  mean number of reads in targeted locus
Quality scores | 1 day
  block and concordance scores, evaluated from 0 to 1 as described in Pacault et al, Plos One, 2023
Optimal window in terms of gestational age for maternal sampling | through study completion, an average of 2 years
  block and concordance scores will be compared depending on the maternal blood sampling window:
  * group 1 corresponds to samples between 7+0 and 7+6 weeks of gestation
  * group 2 corresponds to samples between 8+0 and 8+6 weeks of gestation
  * group 3 corresponds to samples between 9+0 and 9+6 weeks of gestation
  * group 4 corresponds to samples between 10+0 and 10+6 weeks of gestation
  * group 5 corresponds to samples between 11+0 and 11+6 weeks of gestation
  * group 6 corresponds to samples over 12+0 weeks of gestation
Simplicity of implementation | through study completion, an average of 2 years
  will be quoted 1 to 10 (very simple to poor)
Turnaround time | through study completion, an average of 2 years
  will be evaluated in terms of working half-days
Estimated delay for result in standard care diagnosis condition | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Juliette NECTOUX, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Thierry BIENVENU, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Maternité Port-Royal, service de Gynécologie obstétrique, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pacault M, Verebi C, Champion M, Orhant L, Perrier A, Girodon E, Leturcq F, Vidaud D, Ferec C, Bienvenu T, Daveau R, Nectoux J. Non-invasive prenatal diagnosis of single gene disorders with enhanced relative haplotype dosage analysis for diagnostic implementation. PLoS One. 2023 Apr 24;18(4):e0280976. doi: 10.1371/journal.pone.0280976. eCollection 2023. PMID 37093806